CLINICAL TRIAL: NCT01309126
Title: A Phase 3 Open-Label, Randomized, Multicenter Study of Imprime PGG® in Combination With Cetuximab (Erbitux®) in Subjects With Recurrent or Progressive KRAS Wild Type Colorectal Cancer
Brief Title: Study of Imprime PGG® in Combination With Cetuximab in Subjects With Recurrent or Progressive KRAS Wild Type Colorectal Cancer
Acronym: PRIMUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to enrollment challenges resulting from changing treatment patterns in the use of cetuximab, the study has been terminated. No patients remain on study.
Sponsor: HiberCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-CL-PGG-CRC1031
Record Dates: First submitted 2011-02-08; First posted 2011-03-04 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; KRAS Wild Type; Imprime PGG; Cetuximab; Phase 3; Efficacy; Safety; Recurrent or Progressive KRAS Wild Type Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Imprime PGG + cetuximab (Experimental): Biological/Vaccine + Drug
  Interventions: Biological: Imprime PGG + cetuximab
- Arm 2: cetuximab (Active Comparator): Drug
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Biological: Imprime PGG + cetuximab — Imprime PGG: 4 mg/kg and will be administered weekly in each cycle (Weeks 1-6/Days 1, 8, 15, 22, 29, and 36) preceding the administration of cetuximab Cetuximab: initial dose will be 400 mg/m2 on Cycle 1/Day 1 and subsequent doses will be 250 mg/m2, administered weekly in each cycle (Weeks 1-6/Days 1, 8, 15, 22, 29, and 36)
  Other Names: Imprime PGG; Cetuximab (Erbitux)
  Arms: Arm 1: Imprime PGG + cetuximab
Drug: Cetuximab — Cetuximab: initial dose will be 400 mg/m2 on Cycle 1/Day 1 and subsequent doses will be 250 mg/m2, administered weekly in each cycle (Weeks 1-6/Days 1, 8, 15, 22, 29, and 36)
  Other Names: Cetuximab (Erbitux)
  Arms: Arm 2: cetuximab

SUMMARY:
Study BT-CL-PGG-CRC1031 is a Phase 3, open-label, randomized, multi-center study. Qualified subjects, who have KRAS wild type (WT) colorectal cancer will be randomized in a 2:1 ratio to treatment with either Imprime PGG and cetuximab or cetuximab alone. Subjects will be dosed until progression or discontinuation for some other reason. Efficacy will be assessed via Response Evaluation Criteria in Early Tumors 1.1 (RECIST 1.1); computed tomography (CT) scans will be conducted every 6 weeks. Safety, pharmacokinetics (PK), quality of life, and biomarker parameters will also be assessed.

DETAILED DESCRIPTION:
Study BT-CL-PGG-CRC1031 is a Phase 3, open-label, randomized, multi-center study. Qualified subjects, who have KRAS WT colorectal cancer will be randomized in a 2:1 ratio to either:

Arm 1: Imprime PGG and cetuximab or Arm 2: Cetuximab

Approximately 795 subjects will be randomized into the study. Dosing will occur in 6-week cycles. Imprime PGG will be dosed at 4 mg/kg and will be administered weekly in each cycle (Weeks 1-6/Days 1, 8, 15, 22, 29, and 36) preceding the administration of cetuximab (Arm 1 only). The initial cetuximab dose (both arms) will be 400 mg/m2 on Cycle 1/Day 1 and subsequent doses will be 250 mg/m2 administered weekly in each cycle (Weeks 1-6/Days 1, 8, 15, 22, 29, and 36).

Subjects will be dosed until progressive disease (PD) per RECIST 1.1 or discontinuation of study drug for other reasons; e.g., safety. Following completion of the treatment period of the study, subjects will be monitored for survival until death or loss to follow-up. Tumor measurements and determination of tumor responses will be evaluated according to RECIST 1.1. Safety, PK, quality of life, and biomarker parameters will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Is >18 years old;
2. Has recurrent or metastatic carcinoma of the colon or rectum with documented histological or cytological confirmation;
3. Must be KRAS WT;
4. Has measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to RECIST 1.1;
5. Has never received cetuximab or panitumumab, and has not received any treatment for colorectal cancer within 30 days prior to the first dose of study treatment under this protocol;
6. Has an Eastern Cooperative Oncology Group (ECOG) score of 0-1, with a life expectancy of >3 months;
7. Has received at least 2 prior chemotherapeutic regimens for colorectal cancer;
8. Has adequate bone marrow reserve as evidenced by:

   * Absolute neutrophil count ≥1,500/μL
   * Platelets ≥100,000/μL;
9. Has adequate renal function as evidenced by serum creatinine ≤2.5 × the upper limit of normal (ULN) for the reference lab;
10. Has adequate hepatic function as evidenced by:

    * Aspartate aminotransferase ≤3 × ULN for the reference lab (≤5 × ULN for subjects with known hepatic metastases)
    * Alanine aminotransferase ≤3 × ULN for the reference lab (≤5 × ULN for subjects with known hepatic metastases)
    * Bilirubin <1.5 mg/dL or direct bilirubin <1.0 mg/dL
    * Serum Albumin >3.0 gm/dL
11. Has read, understood and signed the informed consent form (ICF) approved by the Independent Review Board/Independent Ethics Committee (IRB/IEC); and
12. If the subject is a woman of childbearing potential or a fertile man, he/she must agree to use an effective form of contraception during the study and for 60 days following the last dose of study drug (an effective form of contraception is abstinence, a hormonal contraceptive, or a double-barrier method).

Exclusion Criteria:

1. Has a known hypersensitivity to cetuximab, murine proteins, or any component of cetuximab;
2. Has a known hypersensitivity to baker's yeast or has an active yeast infection;
3. Has had previous exposure to Betafectin® or Imprime PGG;
4. Has an active, uncontrolled infection;
5. Has known untreated or symptomatic brain metastases;
6. Had a second malignancy within the previous 5 years, except for basal cell carcinoma, cervical intra-epithelial neoplasia or treated prostate cancer with a prostate-specific antigen (PSA) of <2.0 ng/mL;
7. Has known human immunodeficiency virus or acquired immune deficiency syndrome, hepatitis B, hepatitis C, connective tissue disease, or other clinical diagnosis, ongoing or intercurrent illness that in the Investigators opinion should preclude the subject from participation;
8. If female, is pregnant or breast-feeding;
9. Is receiving concurrent standard and/or investigational anti-cancer therapy or has received such therapy within a period of 30 days prior to the first scheduled day of dosing (investigational therapy is defined as treatment for which there is currently no regulatory-authority-approved indication); or
10. Has previously received an organ or progenitor/stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2011-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 18 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 18 months
Rate of complete response (CR) | 18 months
Rate of partial response (PR) | 18 months
Rate of overall response (CR + PR) | 18 months
Safety and tolerability of the dosing regimen as measured by the incidence and severity of adverse events observed in study participants | 18 months
Sparse pharmacokinetic profile of Imprime PGG will be determined to expand current Imprime PGG PK data | 18 months
  Samples for sparse PK will be taken at specified times on Cycle 1/Day 1 in the first 30 available subjects randomized to Arm 1 (Subjects 1-30). Samples will be collected, at multiple times, in the next 60 subjects randomized to Arm 1 who reach Cycle 2/Day 1 of dosing (subjects 31-90). Additionally, any subject after the first 90 subjects (subjects 91-795) who have a screening/baseline calculated creatinine clearance (based on age, weight and serum creatinine) of <60 mL/minute will have sparse PK samples collected.
Change in Quality of Life | 18 months

CONTACTS AND LOCATIONS:
Locations (53):
- United States (44):
  - Northwest Alabama Cancer Center, Florence, Alabama
  - Highlands Oncology Group, Bentonville, Arkansas
  - Pacific Medical Center, Anaheim, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Providence St. Joseph Medical Center, Burbank, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Kenmar Research Institute, Los Angeles, California
  - AMPM Research Clinic, Miami Gardens, Florida
  - MD Anderson Cancer Center, Orlando, Florida
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Indiana University Cancer Center, Beech Grove, Indiana
  - University of Louisville/James Brown Cancer Center, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri- Columbia, Columbia, Missouri
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Hematology and Oncology Associates of Central NY, East Syracuse, New York
  - New York Oncology, Hematology, P.C., Hudson, New York
  - Signal Point Hematology/Oncology, Middletown, Ohio
  - Toledo Community Oncology Program- Toledo Community Hospital, Toledo, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Cancer Centers of the Carolinas, Spartanburg, South Carolina
  - The Jones Clinic, Germantown, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Texas Oncology-Amarillo, Amarillo, Texas
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology Denton South, Denton, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Texas Oncology - Lewisville, Lewisville, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Northern Utah Associates, Ogden, Utah
  - Virginia Oncology Associates, Newport News, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., dba Blue Ridge Cancer Care, Roanoke, Virginia
- Centre d' Oncologie de Gentilly, Nancy, France
- Germany (7):
  - Klinikum Kassel GmbH Medizinische Klinik IV Onkologie, Hämatologie, Immunologie, Kassel, Hessen, Germany
  - Medizinisches Versorgungszentrum Ãrzteforum Seestrabe, Berlin
  - Ãrzteforum Henningsdorf Darmzentrum Oberhavel, Hennigsdorf
  - Universitätsklinikum Köln - Studienzentrum der Klinik I für Innere Medizin, Koeln, Nordrhein Westfalen
  - Schwerpunktpraxis für Hämatologie und Onkologie, Magdeburg
  - Universitaetsklinikum Ulm, Ulm
  - Petruskrankenhaus Wuppertal, Klinik fuer Innere Medizin II- Gastroenterologie, Hepatologie und Diabetologie, Wuppertal
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico